CLINICAL TRIAL: NCT05219448
Title: Reducing Sugared Fruit Drinks in Alaska Native Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Alaska Fairbanks (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Donald Chi, Professor, Oral Health Sciences, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00009185; U01DE027629 (NIH)
Record Dates: First submitted 2022-01-07; First posted 2022-02-02 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Alaska Native; children; sugared fruit drinks; sugar sweetened beverages; oral health; dental
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: There are 2 arms in the study. In Communities A and B, a total of 136 children (and at least one primary caregiver for each child) will be recruited for the intervention and outcomes measured over 12 months. In Community C, 56 children (and at least one primary caregiver for each child) will be recruited to a control group where outcomes are measured over 12 months but the intervention is not delivered until the study data collection period is over.
Who Masked: Outcomes Assessor
Masking Description: All raw data provided to the statistician will include a participant-level variable indicating the community in which the participant lives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and self-efficacy coaching (Experimental): This arm will receive education, behavior change support in the form of self-efficacy coaching, and introduction of sugar-free water enhancers.
  Interventions: Behavioral: Education and self-efficacy coaching
- Comparison (No Intervention): This arm will have the outcomes assessed but will not receive relevant parts of the intervention (education, behavior change support, and introduction of sugar-free water enhancers) until the end of the study.

INTERVENTIONS:
Behavioral: Education and self-efficacy coaching — Children and their caregiver(s) in the intervention communities will receive a culturally-adapted, 5-session program consisting of video-based health education and self-efficacy coaching delivered by an indigenous Community Health Worker. Families will be introduced to sugar-free water enhancers that are commercially available and come in the same flavors as regular Tang and Kool-Aid. The sessions will include conversations on related topics, interactive hands-on activities, and homework assignments. Additionally, four brief "check-ins" will keep families engaged. Local stores in the intervention communities only will carry the sugar-free water enhancers that are highlighted in the health education.
  Arms: Education and self-efficacy coaching

SUMMARY:
This study in Alaska will test whether providing sugar-free alternatives to sugared fruit drinks and introducing education and social support will help families and children to reduce the amount of sugared fruit drinks consumed (measured through the primary outcome of added sugar intake).

DETAILED DESCRIPTION:
Alaska Native children consume an average of 50 teaspoons of sugar per day and most of this added sugar is from fruit drinks like Tang and Kool-Aid. The goal of this community-based behavioral trial is to reduce added sugar intake in Alaska Native children. In Communities A and B, a total of 136 children ages 1-11 years will be recruited for a 6-month culturally-adapted, 5-session intervention consisting of video-based health education and self-efficacy coaching delivered in person by an indigenous Community Health Worker. There will be 4 brief "check-ins" to provide social support. Local stores have been recruited to carry sugar-free fruit drinks. In Community C, 56 children will be recruited to a no treatment control group. Outcomes will be measured at baseline, 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Child must be older than age 1 year but less than age 12 years at time of enrollment. Multiple children from the same family are eligible;
* Child must live in one of the study communities at baseline;
* Child's parent or primary caregiver must of Yup'ik descent, be age 18 years or older, and willing to provide written consent to study procedures;
* Child participant(s) ages 8 to 11 years must be willing to provide written assent to study procedures;
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Severe medical condition that would prevent the child from completing the study procedures;
* Allergy to sucralose or acesulfame potassium (sweeteners in the sugar-free water enhancers) as defined by parent report of any known allergies;
* Sulfa drug allergy (potential hypersensitivity to acesulfame potassium);
* Member of the same household as the Community Health Worker who will be delivering the intervention.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 334 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Chi, DDS, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chi DL, Lewis FM, Weinstein P, Mancl L, Milgrom P, Edwards T, Coldwell S, O'Brien D, Bersamin A, Hopkins S, Orr E, Rivera P, Lenaker D, Sylvetsky A, Gittelsohn J, Walter P, Randall CL, Wiseman D, Dock A, Ko A, Orack J, Nemawarkar D, Panchal S, Soper J, Hill CM, Kerr D, Nguyen DP, Chen CY, MacLachlan E. Healthy Drinks, Healthy Teeth - Ciunerkaq Tanqigtuq (The Future is Bright): A study protocol for a community-based, non-randomized sociobehavioral trial to reduce added sugar intake in Alaska Native Yup'ik children in the Yukon-Kuskokwim Delta. Contemp Clin Trials. 2024 Dec;147:107734. doi: 10.1016/j.cct.2024.107734. Epub 2024 Nov 1. PMID 39489399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by phone and local radio in the communities between 8/26/2022 and 9/16/2022. Participants were screened and enrolled at the community clinics. In the two intervention group communities, 143 children and 81 caregivers were enrolled between 9/6/2022 and 9/13/2022. In the control group community, 58 children and 27 caregivers were enrolled at the community clinic between 9/14/2022 and 9/16/2022. Additional (secondary) caregivers were enrolled at subsequent visits.
Pre-assignment Details: Primary caregivers were enrolled and assigned to units (households). Multiple children could be enrolled from the same household. If the primary caregiver enrolled at baseline was not available, additional (secondary) caregivers were enrolled after baseline.
Units Other Than Participants: Community
Groups:
- Intervention Arm: This arm includes child participants and their caregivers from two communities (intervention community A and intervention community B). The participants in these communities will receive education, behavior change support in the form of self-efficacy coaching, and introduction of sugar-free water enhancers.
  Education and self-efficacy coaching: Children and their caregiver(s) in the intervention communities will receive a culturally-adapted, 5-session program consisting of video-based health education and self-efficacy coaching delivered by an indigenous Community Health Worker. Families will be introduced to sugar-free water enhancers that are commercially available and come in the same flavors as regular Tang and Kool-Aid. The sessions will include conversations on related topics, interactive hands-on activities, and homework assignments. Additionally, four brief "check-ins" will keep families engaged. Local stores in the intervention communities will carry the sugar-free water enhancers that are highlighted in the health education.
- Comparison Arm: This arm includes child participants and their caregivers from one community (community C) and will have the outcomes assessed but will not receive relevant parts of the intervention (education, behavior change support, and introduction of sugar-free water enhancers) until the end of the study.
Period: Overall Study
Arm/Group | Intervention Arm | Comparison Arm
Started | 241; 2 Community (143 children and 77 primary caregivers enrolled at baseline and started the study in the intervention arm. 7 secondary caregivers were enrolled and started at 1-month. 3 secondary caregivers were enrolled and started at 3-months. 5 secondary caregivers were enrolled and started at 6-months. 3 secondary caregivers were enrolled and started at 12-months. Overall, 4 caregivers and 5 children were lost to follow up.) | 93; 1 Community (58 children were enrolled and started the study at baseline. 27 caregivers were enrolled and started the study at baseline. 6 secondary caregivers were enrolled and started the study at 1-month. 2 secondary caregivers were enrolled and started the study at 3-months.)
Baseline | 220; 2 Community (143 children and 81 primary caregivers enrolled at baseline and started the study in the intervention arm.) | 85; 1 Community (58 children and 27 primary caregivers enrolled at baseline and started the study in the comparison arm.)
1-month Data Collection | 231; 2 Community (143 children and 81 primary caregivers were enrolled at baseline and started the study; and 11 secondary caregivers were enrolled at 1-month in the intervention arm.) | 91; 1 Community (58 children and 27 primary caregivers were enrolled at baseline and started the study; and 6 secondary caregivers were enrolled at 1-month in the comparison arm.)
3-month Data Collection | 234; 2 Community (143 children and 81 primary caregivers were enrolled at baseline and started the study; 7 secondary caregivers were enrolled at 1-month in the intervention arm; and 3 secondary caregivers were enrolled at 3-months.) | 93; 1 Community (58 children and 27 primary caregivers were enrolled at baseline and started the study; 6 secondary caregivers were enrolled at 1-month; and 2 secondary caregivers were enrolled at 3-months in the comparison arm.)
6-month Data Collection | 231; 2 Community (143 children and 81 primary caregivers were enrolled at baseline and started the study; 7 secondary caregivers were enrolled at 1-month in the intervention arm; 3 secondary caregivers were enrolled at 3-months; and 4 secondary caregivers were enrolled at 6-months. 4 children and 3 primary caregivers were lost to follow up at this milestone (231 completed 6-months).) | 93; 1 Community (58 children and 27 primary caregivers were enrolled at baseline and started the study; 6 secondary caregivers were enrolled at 1-month; and 2 secondary caregivers were enrolled at 3-months in the comparison arm.)
12-month Data Collection | 232; 2 Community (143 children and 81 primary caregivers were enrolled at baseline and started the study; 7 secondary caregivers were enrolled at 1-month in the intervention arm; 3 secondary caregivers were enrolled at 3-months; and 5 secondary caregivers were enrolled at 6-months. 4 children and 3 primary caregivers were lost to follow up at 6-months. 3 secondary caregivers were enrolled at 12-months. 1 child and 1 primary caregiver were lost to follow up at this milestone (232 completed 12-months)) | 93; 1 Community (58 children and 27 primary caregivers were enrolled at baseline and started the study; 6 secondary caregivers were enrolled at 1-month; and 2 secondary caregivers were enrolled at 3-months in the comparison arm.)
Completed | 232; 2 Community | 93; 1 Community
Not Completed | 9; 0 Community | 0; 0 Community
Not completed — Lost to Follow-up | 9 | 0

BASELINE CHARACTERISTICS:
Population: Children and primary caregivers represent the overall number of baseline participants. Households are also considered as a unit of analysis. Multiple caregivers of child participants were enrolled in some households, but only after baseline. Baseline data was only collected for primary caregivers, so the number of households in each arm by proxy represents the number of caregivers with baseline characteristics analyzed.
Units Other Than Participants: Households (primary caregivers)
Groups:
- Intervention Arm: This arm includes child participants and their caregivers from two communities that will receive education, behavior change support in the form of self-efficacy coaching, and introduction of sugar-free water enhancers.
  Education and self-efficacy coaching: Children and their caregiver(s) in the intervention communities will receive a culturally-adapted, 5-session program consisting of video-based health education and self-efficacy coaching delivered by an indigenous Community Health Worker. Families will be introduced to sugar-free water enhancers that are commercially available and come in the same flavors as regular Tang and Kool-Aid. The sessions will include conversations on related topics, interactive hands-on activities, and homework assignments. Additionally, four brief "check-ins" will keep families engaged. Local stores in the intervention communities will carry the sugar-free water enhancers that are highlighted in the health education.
- Comparison Arm: This arm includes child participants and caregivers from one community that will have the outcomes assessed but will not receive relevant parts of the intervention (education, behavior change support, and introduction of sugar-free water enhancers) until the end of the study.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Comparison Arm | Total
Number analyzed (Participants) | 220 | 85 | 305
Number analyzed (Households (primary caregivers)) | 77 | 27 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] — Child participant age Population: Child participants in the intervention arm at baseline N=143. Child participants in the comparison arm N=58
  years
    number analyzed (Participants) | 143 | 58 | 201
    (all) | 6.1 (2.85) | 6.1 (3.0) | 6.1 (3.0)
Age, Continuous [Mean (Standard Deviation); unit: years] — Primary caregiver age
  years | 37.6 (11.75) | 36.7 (10.4) | 37.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Child participant sex Population: Child participants in intervention arm N=143. Child participants in comparison arm N=58
  Participants
    number analyzed (Participants) | 143 | 58 | 201
    Female | 65 | 24 | 89
    Male | 78 | 34 | 112
Sex: Female, Male [Count of Units; unit: Households (primary caregivers)] — Primary caregiver sex Population: Primary caregivers in intervention arm N=77. Primary caregiver in comparison arm N=27.
  Households (primary caregivers)
    number analyzed (Participants) | 77 | 27 | 104
    Female | 64 | 26 | 90
    Male | 13 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Child participant and primary caregiver race. Alaskan native (Yup'ik) race/ethnicity was part of the inclusion criteria for all participants.
  Participants
    Alaskan Native, Yup'ik | 220 | 85 | 305
Region of Enrollment [Number; unit: participants] — Child participants (N=143) and primary caregivers (N=77) region of enrollment.
  participants
    United States | 220 | 85 | 201
Children in the household [Mean (Standard Deviation); unit: number of children] — The total number of children in each household was measured, including enrolled child participants. Population: Caregivers and children from 77 households in the intervention arm, and 27 households in the control arm were enrolled. Multiple children from the same household could be enrolled.
  number of children
    number analyzed (Participants) | 77 | 27 | 104
    (all) | 3.4 (2.0) | 3.5 (1.3) | 3.4 (1.9)
Household size [Mean (Standard Deviation); unit: people] — The number of people living in each household including children and adults was measured at baseline. Population: Caregivers and children from 77 households in the intervention arm, and 27 households in the control arm were enrolled. Multiple children from the same household could be enrolled.
  people
    number analyzed (Participants) | 77 | 27 | 104
    (all) | 6.4 (2.6) | 6.1 (1.7) | 6.2 (2.6)
Household income [Count of Units; unit: Households (primary caregivers)] — Population: Caregivers and children from 77 households in the intervention arm, and 27 households in the control arm were enrolled.
  Households (primary caregivers)
    number analyzed (Participants) | 77 | 27 | 104
    less than $10,000 | 28 | 6 | 34
    $10,000 to $14,999 | 12 | 2 | 14
    $15,000 to $24,999 | 13 | 4 | 17
    $25,000 to $34,999 | 3 | 4 | 7
    $35,000 to $49,999 | 0 | 1 | 1
    $50,000 to $74,999 | 3 | 4 | 7
    $75,000 to $99,999 | 3 | 1 | 4
    Refused/Did not wish to answer | 15 | 5 | 20
Money for utilities [Count of Units; unit: Households (primary caregivers)] — Responses to this question from primary caregivers were collected at baseline: "How often does money for household utilities (i.e., water, fuel oil, electricity, etc.) run out before the end of the month?" Population: Caregivers and children from 77 households in the intervention arm, and 27 households in the control arm were enrolled.
  Households (primary caregivers)
    number analyzed (Participants) | 77 | 27 | 104
    Never | 24 | 8 | 32
    Seldom | 9 | 4 | 13
    Sometimes | 20 | 12 | 32
    Most times | 14 | 1 | 15
    Always | 6 | 1 | 7
    Refused/Did not wish to answer | 4 | 1 | 5
Traditional Yup'ik Lifestyle [Count of Units; unit: Households (primary caregivers)] — Responses to this question were collected from primary caregivers at baseline: "How much do you follow the traditional Yup'ik way of life?" Population: Caregivers and children from 77 households in the intervention arm, and 27 households in the control arm were enrolled. Multiple children from the same household could be enrolled.
  Households (primary caregivers)
    number analyzed (Participants) | 77 | 27 | 104
    A lot | 53 | 17 | 70
    Sometimes | 24 | 10 | 34
    Rarely | 0 | 0 | 0
    Never | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Added Sugar Intake Among Children
Description: Added sugar intake among children will be measured with a validated hair biomarker, generated from stable carbon and nitrogen isotope ratios of hair using coefficients for added sugar determined specifically for the Yup'ik population. The investigators will measure added sugar in grams of added sugar per day.
Time Frame: Baseline to 6 months
Population: Analysis measuring change in added sugar intake (grams per day) from baseline to 6-months was conducted with available hair biomarker data for children who had hair specimens collected at both events. Out of 143 children with hair samples collected at baseline in the intervention arm, 90 also had hair samples collected at 6-months. Out of 58 children with hair samples collected at baseline in the comparison arm, 38 also had hair samples collected at 6-months.
Measure: Mean (95% Confidence Interval); unit: g/day
Groups:
- Intervention Arm: Children from the intervention community A and community B
- Comparison Arm: Children from the control community C, who did not receive the intervention.
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 90 | 38
g/day | 11.7 [5.7 to 17.7] | 19.1 [10.2 to 28.0]
Statistical Analysis 1: Comparison: Intervention Arm vs Comparison Arm; Null hypothesis: The change in added sugar intake from baseline to 6-months will be the same when compared to children in the no-treatment control arm (measured through hair biomarker); Test type: Superiority; p = 0.17, Regression, Linear — Unadjusted p value presented. The a priori threshold for statistical significance is 0.05; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-3.2 to 18.0]

2. Secondary Outcome: Change in Added Sugar Intake Among Caregivers
Description: Added sugar intake among caregivers will be measured with a validated hair biomarker, generated from stable carbon and nitrogen isotope ratios of hair, based on coefficients for added sugar determined specifically for the Yup'ik population. The investigators will measure added sugar in grams of added sugar per day.
Time Frame: Baseline to 6 months
Population: Analysis measuring change in added sugar intake (grams per day) from baseline to 6-months was conducted with available hair biomarker data for caregivers who had hair specimens collected at both events. Out of 42 caregivers in community A, 35 in community B, and 27 in community C, with hair samples collected at baseline in the intervention arms, 23, 24, and 19 respectively, also had hair samples collected at 6-months.
Measure: Mean (95% Confidence Interval); unit: g/day
Groups:
- Intervention Arm A: Caregivers from the intervention arm community A.
- Intervention Arm B: Caregivers from the intervention arm community B.
- Comparison Arm: Caregivers from the control arm, community C.
Arm/Group | Intervention Arm A | Intervention Arm B | Comparison Arm
Number analyzed (Participants) | 23 | 24 | 19
g/day | 13.6 [1.5 to 25.7] | 33.3 [20.8 to 45.7] | 8.5 [-6.3 to 23.3]
Statistical Analysis 1: Comparison: Intervention Arm A vs Comparison Arm; Null hypothesis: The change in added sugar intake from baseline to 6-months will be the same for caregivers in community A arm when compared to caregivers in the no-treatment control arm (measured through hair biomarker); Test type: Superiority; p = 0.60, Regression, Linear — Unadjusted P-value. The threshold for significance is 0.05; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-24.3 to 14.0]
Statistical Analysis 2: Comparison: Intervention Arm B vs Comparison Arm; Null hypothesis: The change in added sugar intake from baseline to 6-months will be the same for caregivers in community B when compared to caregivers in the no-treatment control arm (measured through hair biomarker); Test type: Superiority; p = 0.013, Regression, Linear — The P-value is unadjusted. The threshold for significance is 0.05; Mean Difference (Final Values) = -24.7, 95% CI 2-sided [-44.1 to -5.4]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from day 3 after baseline (after the sugar-free Kool-aid was introduced), up to the final data collection visit at 12-months.
Description: Adverse events data were collected in two ways throughout the study from day 3 after baseline to 12-months: (1) participants could self-report adverse events to the community health worker they interacted with during study intervention visits; or (2) study staff probed for adverse events during data collection visits at 1-month, 3-months, 6-months and 12-months. Adverse events data were NOT collected in the comparison arm since that arm were not exposed to the sugar-free Kool-aid.
Groups:
- Intervention Arm: Children (N=143) and all caregivers enrolled throughout the duration of the study (N=99) from the intervention arm, where sugar free-Kool aid was introduced in community A and community B. Adverse events data were NOT collected in the comparison arm since that arm were not exposed to the sugar-free Kool-aid.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/242
Serious Adverse Events (participants affected / at risk) | 0/242
Other Adverse Events (participants affected / at risk) | 8/242
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=242)
[child] Upset stomach (possible relation) (Gastrointestinal disorders) | 1 (1) — Child participants reported experiencing mild side-effects of having an upset stomach that they believe was possibly due to consumption or over-consumption of the sugar-free Kool-Aid water enhancers.
[child] Upset stomach (probable relation) (Gastrointestinal disorders) | 2 (2) — Child participants reported experiencing mild side-effects of having an upset stomach that they believe was probably due to consumption or over-consumption of the sugar-free Kool-Aid water enhancers.
[child] Diarrhea (possible relation) (Gastrointestinal disorders) | 2 (2) — Child participants reported experiencing mild side-effects of having diarrhea that they believe was possibly due to consumption or over-consumption of the sugar-free Kool-Aid water enhancers.
[child] Diarrhea (probable relation) (Gastrointestinal disorders) | 2 (3) — Child participants reported experiencing mild side-effects of having diarrhea that they believe was probably due to consumption or over-consumption of the sugar-free Kool-Aid water enhancers.
[caregiver] Diarrhea (probable relation) (Gastrointestinal disorders) | 1 (1) — Adult participants reported experiencing mild side-effects of having diarrhea that they believe was probably due to consumption or over-consumption of the sugar-free Kool-Aid water enhancers.

LIMITATIONS AND CAVEATS:
Allocation was not randomized. Communities were allocated to the intervention arm vs. control arm based on readiness to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05219448/Prot_SAP_ICF_000.pdf